CLINICAL TRIAL: NCT01599819
Title: BAX 855 (PEGylated Recombinant Factor VIII): A Phase 1, Prospective, Open Label, Cross-Over, Dose-Escalation Study in Previously Treated Patients (PTPs) With Severe (FVIII < 1%) Hemophilia A
Brief Title: BAX 855 Dose-Escalation Safety Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Baxter Innovations GmbH (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 261101; 2011-002011-28 (EudraCT Number)
Record Dates: First submitted 2012-05-15; First posted 2012-05-16 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; BAX 855

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): Low dose of ADVATE followed by low dose of BAX 855
  Interventions: Biological: Antihemophilic Factor (Recombinant) - Plasma/Albumin Free Method; Biological: PEGylated Recombinant Factor VIII
- Cohort 2 (Experimental): High dose of ADVATE followed by high dose of BAX 855
  Interventions: Biological: Antihemophilic Factor (Recombinant) - Plasma/Albumin Free Method; Biological: PEGylated Recombinant Factor VIII

INTERVENTIONS:
Biological: Antihemophilic Factor (Recombinant) - Plasma/Albumin Free Method — 1 PK infusion of ADVATE (low dose in Cohort 1, high dose in Cohort 2)
  Other Names: ADVATE
Biological: PEGylated Recombinant Factor VIII — 1 PK infusion of BAX 855 (low dose in Cohort 1, high dose in Cohort 2)
  Other Names: BAX 855

SUMMARY:
The objectives of this study are to assess the tolerability and safety after single dose treatments of BAX 855 in previously treated patients (PTPs) with severe hemophilia A, to determine the pharmacokinetic (PK) parameters of BAX 855 compared in crossover with ADVATE, and to evaluate the impact of anti-polyethylene glycol (PEG) antibodies on PK parameters.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male and is 18 to 65 years of age at the time of screening
* The subject has severe hemophilia A (factor VIII level < 1%)
* The subject was previously treated with plasma-derived factor VIII (FVIII) concentrates or recombinant FVIII for at least 150 exposure days (EDs)

Exclusion Criteria:

* The subject has a detectable FVIII inhibitor at screening, with a titer >= 0.6 BU
* The subject has a documented history of FVIII inhibitors with a titer >= 0.4 BU at any time prior to screening
* The subject has a known hypersensitivity towards mouse or hamster proteins or to polyethylene glycol (PEG)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-09-30 (Actual); Primary Completion 2012-07-27 (Actual); Study Completion 2012-07-27 (Actual)

PRIMARY OUTCOMES:
Serious and non-serious AEs | 4 weeks after infusion with BAX 855 and ADVATE

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (8):
- Specialized Hospital for Active Treatment "Joan Pavel", Sofia, Bulgaria
- Germany (3):
  - Vivantes Klinikum im Friedrichshain, Hemophilia Care Center for Children and Adults, Berlin
  - UKGM Uniklinikum Giessen & Marburg, Giessen
  - Harrison Clinical Research Deutschland, Munich
- Japan (2):
  - Nara Medical University Hospital, Nara
  - Tokyo Medical University Hospital, Tokyo
- United Kingdom (2):
  - Quintiles Drug Research Unit at Guy´s Hospital, London
  - Manchester Haemophilia Comprehensive Care Centre, Manchester Royal Infirmary, Manchester

REFERENCES:
- [Derived] Konkle BA, Stasyshyn O, Chowdary P, Bevan DH, Mant T, Shima M, Engl W, Dyck-Jones J, Fuerlinger M, Patrone L, Ewenstein B, Abbuehl B. Pegylated, full-length, recombinant factor VIII for prophylactic and on-demand treatment of severe hemophilia A. Blood. 2015 Aug 27;126(9):1078-85. doi: 10.1182/blood-2015-03-630897. Epub 2015 Jul 8. PMID 26157075